CLINICAL TRIAL: NCT04364126
Title: Home Blood Pressure Monitoring in Kidney Transplant Recipients to Alleviate Hypertension - a Pragmatic, Registry-based, Randomized Controlled Study
Brief Title: Home Blood Pressure Monitoring in Kidney Transplant Recipients
Acronym: HOBiT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Dag Olav Dahle, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 109164
Record Dates: First submitted 2020-04-22; First posted 2020-04-27 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Hypertension; Cardiovascular Diseases; Kidney Transplant; Complications
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 parallel group study with baseline and follow-up measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (Active Comparator): Clinical blood pressure measured at regular visits
  Interventions: Other: Clinic blood pressure
- Home blood pressure monitoring (Experimental): Home blood pressure measured daily for 1 week before regular clinical visits
  Interventions: Device: Home blood pressure apparatus

INTERVENTIONS:
Device: Home blood pressure apparatus — Target <125/80 mmHg
  Arms: Home blood pressure monitoring
Other: Clinic blood pressure — Target <130/80 mmHg
  Arms: Standard of care

SUMMARY:
Randomized controlled study of home blood pressure monitoring in kidney transplant recipients.

DETAILED DESCRIPTION:
Adult kidney transplant recipients (n=458) will be randomized 1:1 to standard-of-care (SOC) or home blood pressure measurement (HBPM). The SOC group will target office blood pressure <130/80 mmHg. The HBPM group will measure BP at home, twice morning and evening for (3-)7 days before routine clinical visits (ideally 28 measurements); the mean value from day 2-7 is used; target home mean BP is < 125/80 mmHg.

ELIGIBILITY:
Inclusion Criteria:

1. Kidney transplant recipient
2. Male or female subject ≥ 18 years old
3. Any or more of the following at the baseline clinic

   * Conventional office BP ≥130 mmHg systolic and/or ≥ 80 mmHg diastolic
   * HBPM ≥125 mmHg systolic and/or ≥ 80 mmHg diastolic measured within the last 3 months (see appendix 1 for details on methodology)
   * Daytime ambulatory blood pressure monitoring (ABPM) ≥125 mmHg systolic and/or ≥ 80 mmHg diastolic measured within the last 3 months
4. Signed informed consent and expected cooperation of the patient for the treatment and follow up.
5. Have a national personal identification number and not be expected to emigrate during study
6. Enlisted in the Norwegian Renal Registry

Exclusion Criteria:

1. Standing systolic BP < 110 mmHg (to avoid adverse events). Measured after one and three minutes of standing. Not applicable if unable to stand due to wheelchair use.
2. Diagnosed atrial fibrillation (automated monitors not validated)
3. Unwilling to self-monitor
4. Female participant who is pregnant, lactating or planning pregnancy during the trial (management of essential hypertension in pregnancy is different)
5. Arm circumference too large or small to allow accurate BP measurement with available device (22-42 cm).
6. Any reason likely limiting adherence to interventions, as judged by the investigator; examples include active alcohol or substance abuse within the last 12 months, significant poor compliance with medications or attendance at clinic visits, residence in a nursing home, dementia, other medical or psychiatric conditions that may interfere with study participation.
7. Graft- or life expectancy less than 2 years, as judged by the investigator.
8. Current use of ≥ 4 antihypertensive medications
9. More than half of regular appointments planned as remote (e.g. phone or video) consultations.
10. Severe white-coat hypertension, e.g. patients already treated solely based on home BP values.
11. Multi-organ transplants (e.g. heart, lung, liver), though pancreas or beta-cell islet transplant is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Office systolic blood pressure (BP) | 1 year
  As reported to Norwegian Renal Registry

SECONDARY OUTCOMES:
Office diastolic BP | 1 year
  As reported to Norwegian Renal Registry
Proportion with BP below target (office BP <130/80 mmHg) | 1 year
  As reported to Norwegian Renal Registry
Number of BP lowering medications | 1 year
  As reported to Norwegian Renal Registry
Treatment satisfaction | 1 year
  According to study-specific questionnaire in Norwegian. Scores of 1-5, higher scores indicating higher satisfaction.
Concentration of plasma creatinine | 1 year
  As reported to Norwegian Renal Registry
Urine protein/creatinine ratio | 1 year
  As reported to Norwegian Renal Registry

OTHER OUTCOMES:
Number of patients with cardiovascular events | 1 year
  As reported to the Norwegian Renal Registry. Safety endpoint. Includes myocardial infarction, stroke, coronary artery bypass grafting or -angioplasty, other cardiac surgery.
Number of participants with kidney graft loss | 1 year
  As reported to the Norwegian Renal RegistrySafety. Safety endpoint. Includes return to dialysis or re-transplant.
Number of participants with kidney graft rejection | 1 year
  As reported to Norwegian Renal Registry. Safety endpoint.
Number of deaths | 1 year
  As reported to Norwegian Renal Registry. Safety endpoint
Overall quality of life | 1 year
  According to study-specific questionnaire in Norwegian. Scores of 1-5, higher scores indicating higher quality of life.
Hypotensive episodes | 1 year
  According to study-specific questionnaire in Norwegian. Self-reported safety endpoint. Questions about A) Pre-syncope (3 categories: never; a few; montly or more); B) Syncope (3 categories: never; once; multiple). C) If syncope, free text if any trauma was experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Dag Olav Dahle, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Rikshospitalet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No